CLINICAL TRIAL: NCT06039800
Title: Patient Reported Outcome Measures (PROMS): Follow up of Shouldice Hospital Patients
Brief Title: Patient-reported Outcomes for Patients Undergoing Surgery at Shouldice Hospital.
Acronym: PROM project
Status: Recruiting | Type: Observational
Sponsor: Shouldice Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShouldiceH
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Hernia
Keywords: hernia; groin hernia
MeSH Terms: conditions — Hernia; Hernia, Inguinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Background:

Previous publications have highlighted limited data on patient outcomes and experiences at Shouldice Hospital. Existing studies from Europe reported outcomes following Shouldice repair but lacked recent data. The current project seeks to optimize patient care and knowledge through systematic follow-up.

Study Objectives:

Establish a patient-reported outcome measure follow-up program. Evaluate postoperative complication rates. Determine important outcomes to patients. Establish and monitor patient satisfaction with decision-making and hernia repair.

Hypotheses/Research Questions:

Several research questions related to patient motivations, outcomes, knowledge, and satisfaction are posed for investigation.

Potential Risks and Benefits:

No anticipated risks to participants. Participants won't directly benefit but contribute to improving patient care and knowledge.

Study Design:

The study employs a prospective follow-up approach. Surveys are sent at specific intervals (30-40 days, 1-year, 3-years, and 5-years) via email.

Consent forms are included in the email, allowing participants to choose their level of involvement. Data is collected from survey responses, patient charts, and operative notes.

Study Population:

All patients aged 16-90 who underwent hernia surgery at Shouldice Hospital are eligible.

Exclusion criteria:

Lack of an email address. The required sample size is unknown, and this study serves as a pilot.

Data Collection:

Data is collected from surveys, patient charts, and operative notes. Consent is obtained through deferred consent (initial contact via email, with consent forms provided).

Safeguards are in place to protect personal health information.

Duration of Study:

Estimated to take 5-6 years. Recruitment/enrollment: 6-12 months. Follow-up: 5 years from the last enrolled participant. Data analysis and write-up: 5 months.

Overlap with Other Projects:

Concerns about overlap with other studies are addressed, and concurrent participation is allowed. Participants can withdraw at any time.

In summary, this research project aims to gather comprehensive data on hernia surgery outcomes, patient experiences, and satisfaction at Shouldice Hospital through a systematic follow-up approach, contributing to the improvement of patient care and knowledge in this field.

DETAILED DESCRIPTION:
Increasing awareness, research, and publications on patient reported outcomes, patient knowledge, and what matters to patients are being done. There is limited data available in these areas at Shouldice Hospital, leaving potential gaps in knowledge and areas of improvement unidentified. Large scale follow-up on the Shouldice Hospital's postoperative complications.

There are two publications within the last 18 years from Europe reporting outcomes following Shouldice repair with a larger number of enrolled individuals. These publications included 3,888 Shouldice repairs. Bittner et al. (2005) published a Meta-analysis analyzing the postoperative outcome following TAPP/TEP (n=1,830) and Shouldice repair (n=1,773). The authors revealed an infection rate of 0.9%, a hematoma rate of 6.4% (higher than in the laparoscopic group) and a seroma rate of 1.2%. The recurrence rate was 2%. Moreover, a 5.4% rate of chronic pain and a 30-days period until return to work were published. These rates were higher in comparison to endoscopic hernia repair (Bittner et al, 2005). In addition, a German matched-pair registry analysis among 2,115 cases of Shouldice repair took place in 2018. The authors published, that for a selected group of patients (average age: 40 years, a large proportion of women of 30%, a mean BMI value of 24 kg/m2 and a proportion of defect sizes up to 3 cm of over 85%) the Shouldice repair can be used for primary unilateral inguinal hernia repair while achieving an outcome comparable to that of Lichtenstein, TEP and TAPP operations (Kockerling et al, 2018). Malik et al. (2016) provided information on the recurrence rate (age-standardized recurrence risk of 1.15%; n=65,148) of patients who were operated on in the Shouldice repair at the Shouldice hospital. But in terms of SSI, SSO and postoperative outcome in general no current information from our Shouldice hospital has been revealed within the last two decades (Malik et al, 2016).

In order to further optimize, evaluate, and increase knowledge of the Shouldice repair systematic follow-up of patients who were operated on at the Shouldice Hospital should be updated. The current project aims to perform a systematic follow-up of patients for the purpose of supporting the ongoing improvement of patient care and knowledge. This study will act as a pilot for refining our long term follow up, focused on patient and surgical outcomes.

Study Objectives:

1. Establish a patient reported outcome measure follow up program at Shouldice Hospital
2. Evaluate the postoperative complication rate (pain, infection, recurrence, and other complications)
3. Determine the reasoning and important outcomes to patients who undergo hernia repair at Shouldice Hospital.
4. Establish and monitor patient satisfaction with decision making and hernia repair.

Hypothesis/Research Questions:

1. What were the most common reasons for patients to undergo hernia repair?
2. What was the most reported important outcome to patients after hernia surgery?
3. Did patients feel they had adequate knowledge and feel a part of the decision-making process?
4. How satisfied and confident were patients with their Shouldice hernia repair at 1-year after surgery?
5. Was there any improvement in quality of life due to hernia repair noted at 1-year after surgery?
6. What is the infection rate, pain incidence, and hernia recurrence rate at 30-days after hernia repair at Shouldice Hospital?
7. What is the pain incidence and hernia recurrence rate at 1-, 3-, and 5-years after hernia repair at Shouldice Hospital?
8. Is there a difference in pain experienced after surgery by patients based off the hernia they had repaired?
9. Does infection rate differ depending on hernia and/or hernia repair?
10. Does infection rate differ for those given or not given antibiotics prior to or during surgery?

Potential Risks and Benefits:

There are no known or anticipated risks to participants as individuals or as part of an identifiable group. This includes no physical, psychological, or emotional, social, and/or data security breach risks. The use of information will remove any personal identifiers before data analysis. There are no direct benefits to the participants from their involvement in the project and these include no education about research methods or useful knowledge about self.

Study Design:

The current study is a prospective follow up of patients who had an operation for a hernia at the Shouldice Hospital. The study design includes using an automated report generated for follow up which will allow for participant identification and provide necessary information to send the consent forms and follow up to patients, as well as responses from follow up surveys by email, and manual review of charts and operative notes. All patients that had surgery at Shouldice Hospital are included unless they did not have an email address. The reason for this exclusion is due to the electronic and internet-based nature of the project. Patients will be emailed 30-40 days after surgery, as well as 1-year, 3-years, and 5-years after surgery using the Hospital's current survey site: Simple Survey. Each email will have a link to a consent form, which will provide potential participants with the choice to be taken directly to the survey if they have consented, decline to participate, or be provided with information to contact a research team member. Patients that do not respond after the 30-40-day postoperative survey will be contacted by phone; this is to ensure comprehensive data collection regarding infection at 30-40 days after surgery. Patients that respond yes to infection questions at the 30-40-day postoperative survey will additionally be asked if we can contact them via telephone to follow up on their potential infection.

The survey is designed to capture the results of important questions and aims about this study. The 30-40 day and 1-year postoperative survey includes a postoperative recovery, preoperative decisions and hernia repair, and final questions and comments section. The 3- and 5-year postoperative surveys have the postoperative recovery and final questions and comments sections. The postoperative recovery portion includes questions regarding pain and swelling (30-40 day/1-year/3-year/5-year survey) from HerniaMed (Stechemesser et al, 2012), questions regarding infection, fluid formation, and hematoma pertaining to grade of surgical site infection and surgical site occurrence (30-40 day survey), and additional questions regarding hernia relapse (30-40 day/1-year/3-year/5-year survey) and wound complication (30-40 day survey). Another part of the survey pertains to preoperative decisions and hernia repair. The 30-40-day postoperative survey enquires about the reasons for surgery, which was used for our purposes of analyzing the reason for having surgery but tailored from Smith et al (2022). This paper by Smith et al (2022) found five superordinate themes when studying what matters to abdominal wall hernia patients, which included body image, mental health, symptoms, interpersonal relationships, and employment. After these questions, patients are asked what the most important outcome was to them after surgery. This question is asked on the 30-40-day postoperative survey and may hold some hindsight bias, but we felt it was important that our ongoing research include these types of questions as patient's responses may differ from the current documented reasons for surgery and important outcomes. Additional questions on the 30-40-day postoperative survey was asked on the knowledge patients had regarding hernia surgery and recovery and how patients felt about being a part of the decision-making process. After reading Rossello Jimenez et al (2022) paper, which was done to understand patient knowledge of hernia surgery (self-reported), we decided that the other variables, when trying to understand important patient perspectives for patient reported outcomes, included if patients had adequate knowledge regarding surgery and recovery as well as if they felt a part of the decision-making team. The preoperative decisions and hernia repair section differs on the 1-year postoperative survey. At the 1-year postoperative time the survey asks patients questions about satisfaction with hernia repair, outcome of hernia repair, and improvement of quality of life with hernia repair. These questions were adapted from the hernia quality of life assessment instrument (HERQL) (Huang et al, 2017). The final part of the surveys allow for further context to patients attitudes towards the Hospital, any major life events that may affect recovery, and additional space for comments.

Study Population:

The population will focus on all patients aged 16-90 years of age, standard age of patients accepted for surgery at Shouldice Hospital, who had a hernia operation at Shouldice Hospital. The only exclusion criteria are those without an email address. The reason for this exclusion is due to the electronic and internet-based nature of the project. As this is the first study of its kind at Shouldice Hospital the required sample size is unknown, and this study will act as an initial pilot for systematic follow up focused on patient and surgical outcomes. However, for the infection rate analysis we know that to compare to the publications on Shouldice Repair in Europe that were written within the last two decades, which had 3,888 individuals combined (Bittner et al. 2005, n=1773; Köckerling et al. 2018, n=2115), we will aim to analyze information from 2,000 patients to allow for a meaningful scientific comparison with current knowledge. Therefore, we aim to contact 4,500 patients in order to analyze a total of 2,000 patients. This is based off information gathered by this institution from previously done prospective projects. When initial research contact was emailed, there was a response rate of 45%. No dropout rate has been measured as we will gather data for this study to go on with a sample size calculation in the future.

Data Collection:

This study will use recorded sources (responses to surveys, patient charts, and operative notes) to collect information. This will include a research team member manually checking patient charts and operative notes as well as downloading and inputting survey responses. Surveys are sent at 30-40 days, 1-year, 3-year, and 5-year postoperative time. Provided in supplemental material is a list of the data we will be collecting to use in data analysis and during the explanations of results.

A study personnel will identify potential study participants through a report that is generated daily, using the hospital database, which is sent and stored as an excel file on the hospitals secure network (EDrive). Only research team personnel will have access to these excel files. The report shows patient Hospital account number, patient first and last name, discharge date, length of hospital stay, patient email address, as well as patient information (sex, smoker, height, and weight). The automated report will be used by a study personnel to upload and send surveys, utilizing SimpleSurvey, at the postoperative times. The contacting person will not be already known to potential participants when making initial contact, however, the potential participants will be known to Shouldice Hospital as they will have had an operation here.

For the purposes of this research project, composed of simple review of charts and operative notes as well as follow up for patient reported outcomes, a consent alteration is requested (deferred consent). As the request for altered consent pertains to TCPS2 3.7A this research project presents as no more than minimal risk to the participants, an alteration to the consent requirement is unlikely to adversely affect the welfare of participants, and it may be impractical (Government of Canada, 2018) to carry out a large scale follow up initiative without an altered consent process. The altered consent process would compromise of deferred consent so that initial contact to send consent forms can be achieved. In person consenting would be impractical as the current hospital procedures for patient intake and during hospital stay would be onerous to other departments as well as a burden to the small number of research department staff. In regard to TCPS2 3.7B each postoperative contact email will immediately notify potential participants of the research project and will have a link to the consent form to ensure consent is obtained and ongoing. On each of the consent forms potential participants will have the choice to be taken directly to the survey if they have consented, decline to take part, or be provided with information to contact a research team member. Potential participants can take as long as they want to decide about participation, but the nature of the study focuses on data collection at specific postoperative intervals. This research is not being done under medical emergencies or involving those with diminished decision-making capacity (TCPS2 3.8-3.11). In regard to PHIPA, this research project will be submitted to an ethics board and researchers will comply with the outlined compliance in section 44. In order to ensure potential participants meet the criteria for follow up (have an email address) and to send a consent form, we require personal information without direct consent, but will obtain consent prior to the collection of all additional information which was not provided in the automated report. Potential participants will be informed about the opportunity to withdraw at any time. By doing so potential participants can refuse to participate or request additional contact/information by research personnel. Steps are taken to safeguard personal health information by password protection and safe storage.

Overlap with other projects is a concern as we aim to have multiple studies running. However, there will be additional populations under review in this project (all hernia types and recurrences) and this project is specifically aimed to pilot a systemic follow up program. Standard follow up procedures and concurrent research participation can be routine practices. Participants will be able to withdraw from participation at any time as well as decline to participate.

Duration of Study:

The study is estimated to take 5-6 years from the beginning of data collection until finishing the write up of results. Recruitment/enrollment will take 6-12 months, follow up will take 5 years from last enrolled participant, and data analysis and study write up will take 5 months. The time it takes for publication is not taken into consideration. Duration of participant participation is dependent on which and how many follow up surveys are completed. It is estimated to take 5 minutes for consent form review (multiplied by 4 consent forms), 3-5 minutes for the 30-40 day postoperative survey, 3 minutes for the 1-year postoperative survey, and 4 minutes for 3- and 5-year postoperative surveys (2 minutes each). The surveys are sent to patients 30-40 days, 1-year, 3-years, and 5-years after surgery. There will only be a follow up phone call reminder for those who don't complete and respond yes to being contacted in regard to the infection questions at the 30-40 day postoperative survey.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 16-90 who underwent hernia surgery at Shouldice Hospital are eligible.

Exclusion Criteria:

* Lack of an email address.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all patients aged 16-90 who underwent hernia surgery at Shouldice Hospital, with the only exclusion being those without an email address. This exclusion is due to the electronic nature of the project. Since this is the first study of its kind at Shouldice Hospital, the required sample size is unknown, and this project serves as a pilot for systematic follow-up on patient and surgical outcomes.
  For the specific analysis of infection rates, the study aims to gather data from 2,000 patients. To achieve this, the researchers plan to contact 4,500 patients, based on information from previous projects. Initial research contact yielded a 45% response rate, and no dropout rate has been measured yet, as data collection for this study will inform future sample size calculations.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence after hernia repair | Recurrence after hernia repair after one year
  Recurrence after hernia repair

SECONDARY OUTCOMES:
Recurrence after hernia repair | Recurrence after hernia repair after three years
  Recurrence after hernia repair
Recurrence after hernia repair | Recurrence after hernia repair after five years
  Recurrence after hernia repair
Recurrence after hernia repair | Recurrence after hernia repair after 30 days
  Recurrence after hernia repair

CONTACTS AND LOCATIONS:
Locations (1):
- Shouldice Hospital, Thornhill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No